CLINICAL TRIAL: NCT00003312
Title: Phase II Trial of Transrectal Ultrasound Guided Permanent Radioactive Implantation of the Prostate for Definitive Management of Localized Adenocarcinoma of the Prostate
Brief Title: Brachytherapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RTOG-9805; CDR0000066259
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Iodine-125

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: iodine I 125

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy through seeds implanted into the prostate may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of brachytherapy in treating patients with stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effectiveness of transrectal ultrasound guided permanent radioactive implantation of the prostate in patients with confined adenocarcinoma of the prostate. II. Assess the overall survival, disease specific survival, clinical relapse (local or distant), PSA levels, and genitourinary and gastrointestinal morbidity in these implant patients. III. Assess the quality of life of these patients.

OUTLINE: This is a multicenter study. Patients receive transrectal ultrasound guided radioactive I-125 seeds implanted into the prostate. At least one week prior to implant, patients undergo transurethral ultrasound study to determine the volume of prostate. Following implantation, seeds that have extruded into the bladder or lodged in the urethral wall are retrieved, and extra seeds may be implanted into identified "cold spots" for uniform seed distribution. Prostate rebiopsy is required before starting hormonal therapy for local progression or biochemical failure without clear focus of progression. Quality of life is assessed every 3 months for 1 year, then every 6 months for 1 year, and then annually for 3 years. Patients are followed every 3 months for 1 year, then every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 95 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locally confined adenocarcinoma of the prostate Stage I or II (T1b-c or T2a-b, NX, M0) PSA no greater than 10 ng/mL Prostate volume by transurethral ultrasound no greater than 45/mm3 at least 1 week, but no more than 4 weeks, prior to implant Gleason score no greater than 6 American Urological Association voiding symptom score no greater than 12 No evidence of distant metastases No lymph node involvement

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No prior or concurrent malignancy within 5 years except basal or squamous cell skin cancer No major medical or psychiatric illness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No prior hormonal therapy, including finasteride Radiotherapy: No prior pelvic radiotherapy Surgery: No prior radical surgery for prostate cancer (e.g., transurethral prostatectomy) No hip prosthesis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 1998-09; Primary Completion 2004-01 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A. Lawton, MD, Study Chair — Medical College of Wisconsin
Locations (258):
- United States (241):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Urology Associates - Mobile AL, Mobile, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscallosa, Alabama
  - Providence Cancer Therapy Center, Anchorage, Alaska
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Cancer Care Center, Pomona, California
  - Mercy Medical Center - Redding, Redding, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - Santa Cruz Radiation Oncology Medical Group, Inc., Santa Cruz, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Radiation Oncology Center - Walnut Creek, Walnut Creek, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Whittingham Cancer Center, Norwalk, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - West Florida Cancer Institute - Pensacola, Pensacola, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - St. Joseph's Radiation Oncology Center, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medical Center at Bowling Green, Bowling Green, Kentucky
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Western Baptist Hospital, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Joint Center for Radiation Therapy, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Regional Medical Center, Midland, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Veterans Affairs Medical Center - Saint Louis, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Elizabeth General Medical Center - West, Elizabeth, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology, P.C., Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - Genesee Hospital - Rochester, Rochester, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Catawba Memorial Hospital, Hickory, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - UNI-MED Medical Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Samaritan Regional Cancer Center, Corvallis, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Penn State Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Catholic Medical Center, Mercy Fitzgerald Divison, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - East Texas Medical Center - Cancer Institute, Tyler, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Virginia Baptist Hospital, Lynchburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Oncology Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (17):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Gillin MT, Dunning BF, Lawton CA, Foley WD, Byhardt RW, Morton G, Baikadi M, Pisansky TT, Michalski JM, Ibbott G, Lopez F; Radiation Therapy Oncology Group. Quality assurance methods for the first Radiation Therapy Oncology Group permanent prostate implant protocol. Brachytherapy. 2006 Jul-Sep;5(3):152-6. doi: 10.1016/j.brachy.2006.05.004. PMID 16864066
- [Result] Lawton CA, Hunt D, Lee WR, Gomella L, Grignon D, Gillin M, Morton G, Pisansky TM, Sandler H. Long-term results of a phase II trial of ultrasound-guided radioactive implantation of the prostate for definitive management of localized adenocarcinoma of the prostate (RTOG 98-05). Int J Radiat Oncol Biol Phys. 2011 Sep 1;81(1):1-7. doi: 10.1016/j.ijrobp.2010.05.056. Epub 2011 Apr 4. PMID 21470793
- [Result] Lawton CA, DeSilvio M, Lee WR, Gomella L, Grignon D, Gillin M, Morton G, Pisansky T, Sandler H. Results of a phase II trial of transrectal ultrasound-guided permanent radioactive implantation of the prostate for definitive management of localized adenocarcinoma of the prostate (radiation therapy oncology group 98-05). Int J Radiat Oncol Biol Phys. 2007 Jan 1;67(1):39-47. doi: 10.1016/j.ijrobp.2006.08.016. Epub 2006 Nov 2. PMID 17084551
- [Result] Feigenberg SJ, Lee WR, Desilvio ML, Winter K, Pisansky TM, Bruner DW, Lawton C, Morton G, Baikadi M, Sandler H. Health-related quality of life in men receiving prostate brachytherapy on RTOG 98-05. Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):956-64. doi: 10.1016/j.ijrobp.2004.12.061. PMID 15989995
- [Result] Lawton CA, DeSilvio M, Lee WR, et al.: Correlating prostate seed implant quality with clinical outcomes for patients treated on RTOG protocol 98-05 (a multi-institutional phase II trial of transrectal ultrasound guided prostate seed implant for localized prostate cancer). [Abstract] American Society of Clinical Oncology 2005 Prostate Cancer Symposium, 17-19 February 2005, Orlando, Florida. A-90, 2005.